CLINICAL TRIAL: NCT06344286
Title: The Effects of Minimal Enteral Nutrition on Mesenteric Blood Flow and Oxygenation Among Neonates With Hypoxic-ischemic Encephalopathy Under Therapeutic Hypothermia
Brief Title: The Effects of Minimal Enteral Nutrition on Mesenteric Blood Flow and Oxygenation in Neonates With HIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, DİDEM ARMAN, Associate Professor, Istanbul Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IstanbulTRH-DArman-002
Record Dates: First submitted 2024-03-12; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Hypoxic-Ischemic Encephalopathy
Keywords: Therapeutic hypothermia; Minimal enteral nutrition; Mesenteric oxygenation; Mesenteric blood flow; Splanchnic oxygenation; Cerebrosplanchnic ratio
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Intervention Model Description: An enteral intake of breast milk with a volume of 10-20 mL/kg/day was defined as minimal enteral feeding. Minimal enteral feeding was initiated at postnatal 24 hours with breast milk via an orogastric tube. A total daily intake of 120 ml/kg/day was defined as full enteral feeding.
  The babies were randomized into two groups based on whether they received MEN during TH. While the babies fed with MEN during TH constituted the study group, the control group was composed of the babies who were given the same amount of distilled water according to the same protocol. Two groups were compared in terms of demographic characteristics, clinical outcomes, NIRS and Doppler measurements.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The feeding materials were prepared inside an opaque syringe and serially numbered by Total Parenteral Nutrition Department in our institution. The investigators who made all measurements, examinations and collected data, and the nurses of the babies were blinded. All of the infants in the study group were fed with breast milk during the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infants receiving MEN (Active Comparator): The babies fed with minimal enteral nutrition during TH constituted the study group
  Interventions: Dietary Supplement: Minimal enteral nutrition
- Infants receiving placebo (Placebo Comparator): The babies who were given distilled water during TH
  Interventions: Dietary Supplement: Distilled water

INTERVENTIONS:
Dietary Supplement: Minimal enteral nutrition — The babies were randomized into two groups based on whether they received MEN during TH. While the babies fed with MEN during TH constituted the study group, the control group was composed of the babies who were given the same amount of distilled water according to the same protocol. Two groups were compared in terms of demographic characteristics, clinical outcomes, NIRS and Doppler measurements.
  Arms: Infants receiving MEN
Dietary Supplement: Distilled water — The babies were randomized into two groups based on whether they received MEN during TH. While the babies fed with MEN during TH constituted the study group, the control group was composed of the babies who were given the same amount of distilled water according to the same protocol. Two groups were compared in terms of demographic characteristics, clinical outcomes, NIRS and Doppler measurements.
  Arms: Infants receiving placebo

SUMMARY:
The goal of this clinical trial is to evaluate the effects of minimal enteral nutrition (MEN) on mesenteric blood flow and oxygenation with Doppler USG and Near Infrared Spectroscopy (NIRS) during therapeutic hypo¬thermia (TH) in babies with hypoxic ischemic encephalopathy. The main question it aims to answer is:

1- How do the mesenteric blood flow and oxygenation get affected with MEN during TH? Participants will be either fed with MEN during TH or given placebo.

DETAILED DESCRIPTION:
Objectives: The investigators aimed to evaluate the effects of minimal enteral nutrition (MEN) on mesenteric blood flow and oxygenation with Doppler USG and Near Infrared Spectroscopy (NIRS) during therapeutic hypo¬thermia (TH) in babies with HIE.

Methods: This prospective, randomized controlled study was conducted between September 2020 to August 2022. The infants receiving MEN during hypothermia (n =30) and those who were not fed (n=30) constituted the study and control groups. Infants were monitored continuously with NIRS and mesenteric arterial blood flow velocities were measured with Doppler USG before and after feeding.

ELIGIBILITY:
Inclusion Criteria:

* The neonates with evidence of encephalopathy de¬fined by seizures or abnormalities on a modified Sarnat exam were enrolled. The hypoxic-ischemic injury was defined by 1. a pH of ≤ 7.0 and/or 2. base deficit >-16 mmol/L recorded in cord blood or blood gas obtained within the first hour postnatally or a pH of 7.0 - 7.15 and/or base deficit (-10-15.9) mmol/L with the presence of an acute perinatal event (cord prolapse, placental abruption, heart rate decelerations, severe fetal bradycardia). In cases where criteria 1 or 2 are met, with the presence of seizures or a diagnosis of moderate to severe encephalopathy according to the Sarnat & Sarnat classification based on neurological examination were treated with TH.

Exclusion Criteria:

* Infants with congenital malformation or hereditary metabolic diseases, infants whose enteral feeding was initiated before randomization and infants without lack of parental consent were excluded. The maternal and neonatal demographic characteristics and clinical outcomes were collected from medical records.

Ages: 0 Days to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Cerebral and mesenteric blood flow velocities and oxygenation | (From postnatal first day until postnatal 4 th day)Doppler US of SMA and MCA performed before feeding (15-30 minutes before) and 60 minutes after feeding
  Cerebral and mesenteric blood flow velocities with Doppler US
Cerebral and mesenteric rSO2 values | (From postnatal first day until postnatal 4 th day) Recording of NIRS data was commenced 60minutes before the initiation of TH and was continued during the procedure till 24 hours after cessation of TH
  Cerebral and mesenteric rSO2 values with NIRS

SECONDARY OUTCOMES:
Development of NEC | From admission to NICU till postnatal 15th day or hospital discharge whichever came first,
  The infants will be monitorized for NEC development
Feeding intolerance | From admission to NICU till postnatal 15th day or hospital discharge whichever came first,
  The infants will be monitorized for feeding intolerance
Time to full enteral feeding | From admission to NICU till postnatal 15th day or hospital discharge whichever came first,
  The infants will be monitorized for the time to full enteral feeding.

CONTACTS AND LOCATIONS:
Overall Officials: DİDEM ARMAN, Principal Investigator — Istanbul Training and Research Hospital
Locations (1):
- IstanbulTRH, Istanbul, Turkey (Türkiye)